CLINICAL TRIAL: NCT00325273
Title: Prevention Allergic Disease of Infant With Probiotics During Pregnancy and Neonate
Brief Title: Prevention Allergic Disease of Infant With Probiotics During Pregnancy and Neonatal Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Chiayu Ou/chief in department of Obstetrics, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: CMRPG84025
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2011-06

CONDITIONS: Atopic Dermatitis; Allergic Rhinitis; Asthma
Keywords: Lactobacillus rhamnosus; Atopic dermatitis; Allergic rhinitis; Asthma; Infant; Pregnancy
MeSH Terms: conditions — Dermatitis, Atopic; Rhinitis, Allergic; Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- probiotics & allergy (Experimental): 1. To understand the preventive effect of probiotics in neonatal peroid
  2. To investate the possible mechanism
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG — use Lactobacillus rhamnosus GG in pregnant women from gestational 26 weeks till newborn 6 months
  Other Names: Brand names: Culturelle DS, Culturelle HS

SUMMARY:
The purpose of this study is to determine whether childhood atopic disease decrease or not after allowing allergic mothers intake of probiotic (Lactobacillus GG) in second trimester, followed by infant intake for 6 months after birth.

DETAILED DESCRIPTION:
The prevalence of atopy at Taiwan increased 8 times in past 20 years and also increased all over the world. In our previous study, maternal atopic history rather than paternal one is the major factor to effect infant eczema and IgE titers. This may be related to maternal inheritance and environments during pregnancy. Kalliomaki et al. (Lancet, vol.357, p1076-9, 2001) presented that Lactobacillus GG used 2-4 weeks prenatally to mothers and 6 months postnatally to infants was effective in prevention of early atopic disease in children at high risk.

We designed a double-blind randomized placebo-controlled study to evaluate whether cord blood IgE and childhood atopic disease decreased after allowing allergic mothers intake of Lactobacillus GG in second trimester, followed by infant intake of Lactobacillus GG for 6 months after birth.

Materials and Methods:

1. Inclusion criteria: Pregnant women with atopic disease, which was determined with atopic history, elevated total IgE > 100 kU/l and positive specific IgE.
2. Case number: 100 cases were collected in both control and study groups.
3. Study design: In a double blind randomized placebo-controlled study, eligible cases are allowed to take Lactobacillus GG or placebo daily from gestational age of 24 weeks until delivery in both groups.

   In study group, Lactobacillus GG is given prenatally from gestational age of 24 weeks to delivery for mothers and 6 months postnatally for infants.

   In control group, placebo starch is given prenatally from gestational age of 24 weeks for mothers to delivery and 6 months postnatally for infants.
4. Schedule of follow-up: Infant/child clinical symptoms and sign are evaluated and IgE and specific IgE are tested in bloods from umbilical cords, infants in 1, 3 and 5 year old.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with atopic disease, which was determined with atopic history, elevated total IgE > 100 kU/l and positive specific IgE

Exclusion Criteria:

* Multiple pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-04; Primary Completion 2008-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of atopic disease in infant | two years

CONTACTS AND LOCATIONS:
Overall Officials: Chia-yu Ou, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Niao-Sung, Taiwan

REFERENCES:
- [Background] Kalliomaki M, Salminen S, Arvilommi H, Kero P, Koskinen P, Isolauri E. Probiotics in primary prevention of atopic disease: a randomised placebo-controlled trial. Lancet. 2001 Apr 7;357(9262):1076-9. doi: 10.1016/S0140-6736(00)04259-8. PMID 11297958
- [Background] Kalliomaki M, Salminen S, Poussa T, Arvilommi H, Isolauri E. Probiotics and prevention of atopic disease: 4-year follow-up of a randomised placebo-controlled trial. Lancet. 2003 May 31;361(9372):1869-71. doi: 10.1016/S0140-6736(03)13490-3. PMID 12788576
- [Derived] Ou CY, Kuo HC, Wang L, Hsu TY, Chuang H, Liu CA, Chang JC, Yu HR, Yang KD. Prenatal and postnatal probiotics reduces maternal but not childhood allergic diseases: a randomized, double-blind, placebo-controlled trial. Clin Exp Allergy. 2012 Sep;42(9):1386-96. doi: 10.1111/j.1365-2222.2012.04037.x. PMID 22925325